CLINICAL TRIAL: NCT00662753
Title: A Structured Program for Hypertension Control in Community Clinics: A Randomized Trial
Brief Title: A Study in the Use of Home Blood Pressure Monitoring and Telephone Follow-up to Control Blood Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP01
Record Dates: First submitted 2008-04-15; First posted 2008-04-21 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2008-04

CONDITIONS: Hypertension
Keywords: hypertension; home blood pressure monitoring; nurse telephone follow up; medically underserved populations
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- home monitoring (Active Comparator): home blood pressure monitor
  Interventions: Device: Home monitoring
- monitor & phone call (Experimental): home blood pressure monitor + phone calls
  Interventions: Other: monitor & phone call

INTERVENTIONS:
Device: Home monitoring — Participants will receive a home blood pressure monitor and be taught how to use it. They will have an education session to review treatment goals, medications, diet and exercise. They will be asked to see their primary care provider at least every 3 months and the research nurse at 3, 6 and 12 months.
  Arms: home monitoring
Other: monitor & phone call — Participants will receive all of the same interventions of the home monitoring group plus they will receive scheduled telephone follow up by the research nurse
  Arms: monitor & phone call

SUMMARY:
The purpose of this study is to determine if the use of home blood pressure monitors plus nurse telephone monitoring is more effective than the use of blood pressure monitors alone in improving control of high blood pressure in an urban medical clinic.

DETAILED DESCRIPTION:
Participants will all have home blood pressure monitors, education session on controlling their blood pressure and will be randomized to recieve 6 months of intensive telephonic on a set monitoring schedule or no telephonic follow up. Phone calls will be weekly for 4 weeks, then every 2 weeks for 8 weeks then monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with essential hypertension
* systolic blood pressure >140 mm Hg (130 if diabetic) OR diastolic blood pressure > 90 mm Hg (80 if diabetic)on at least 2 clinic visits prior to randomization
* BP at time of screening is > than systolic 140 (130 if diabetic) or diastolic 90 (80 if diabetic)
* patient is prescribed at least 1 antihypertensive medication
* Patient is fluent in English
* Patient is easily accessible by telephone

Exclusion Criteria:

* persons with stage 4 or 5 chronic kidney disease or end stage renal disease on dialysis
* Patients with a terminal illness
* Patients with severe dementia or serious mental illness
* Inability to preform self blood pressure monitoring
* Patient lacks a functioning home phone or personal cellular phone
* Pregnant or planning to get pregnant
* Arm circumference exceeds the allowable limit on the largest home BP monitor cuff

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | at 6 mo and 12 mo after randomization

SECONDARY OUTCOMES:
Blood pressure measured at home | 6 and 12 months post randomization
Compliance with use of home blood pressure monitor | 6 and 12 months post randomization
Number and type of antihypertensives prescribed | 12 months post randomization
Patient satisfaction and Quality of Life | 6 and 12 months post randomization
Primary care provider satisfaction with intervention | 6 mo post randomization of a provider's first patient to enroll in the trial
Number of primary care provider visits | 12 months post randomization
Number and quality of adverse events | 3, 6, and 12 months post randomization
cost analysis | 12 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Samir Patel, MD, Principal Investigator — The George Washington University Medical Faculty Associates; Richard Katz, MD, Principal Investigator — The George Washington University Medical Faculty Associates
Locations (2):
- United States (2):
  - Brentwood Unity Health Care Center, Washington D.C., District of Columbia
  - Congress Heights Unity Health Care Center, Washington D.C., District of Columbia